CLINICAL TRIAL: NCT03522623
Title: Estimating Indirect and OOP Costs in Pediatric Inflammatory Bowel Disease: a National Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: University of Ottawa (Other); University of Toronto (Other); University of Alberta (Other); University of Calgary (Other); Dalhousie University (Other); Provincial Health Services Authority British Columbia (Other)
Responsible Party: Principal Investigator, Wael El-Matary, Associate Professor and Section Head, Pediatric GI, University of Manitoba
Other Study IDs: HS20851(H2017:189)
Record Dates: First submitted 2017-11-08; First posted 2018-05-11 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: IBD
Keywords: colitis; costs; Crohn; IBD
MeSH Terms: conditions — Colitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IBD: Children and families with IBD will be surveyed
  Interventions: Other: Non-interventional study

INTERVENTIONS:
Other: Non-interventional study — Non-interventional study

SUMMARY:
inflammation of the gastrointestinal tract. A recent Canadian study from found that Canada has amongst highest incidence rates of childhood-onset IBD (10 per 100,000 for children <16y). In 2012, Crohn's and Colitis Canada estimated that direct medical costs of IBD in Canada were >$1 billion, and estimated indirect costs amounting to $1.8 billion. An American study demonstrated the direct costs of caring for children with IBD was double those for adults. Indirect health care costs in children with IBD have not been well-described. The Canadian Gastro-Intestinal Epidemiology Consortium (CanGIEC) is a pan-Canadian network of new and established IBD clinician-researchers and methodologists from 6 provinces experienced in the use of health administrative data. CanGIEC is evaluating variation in care of children with IBD, and will expand this research stream to assess direct and indirect cost of care. This will involve a collaboration with the CIHR/CHILD Foundation Canadian Children IBD Network (CIDsCaNN), which comprises an inception cohort of children diagnosed at all 12 pediatric IBD centres across Canada.

Hypothesis: Direct health costs are dominated by medication expenses (particularly biologics), with resulting variation within and across provinces in costs and out-of-pocket expenses to the families due to coverage disparity. Indirect costs include school and parental absenteeism, and productivity losses.

Aims:

1. Determine the cost of care of children with IBD, incurred by caregivers,across Canada. Costs include:

   a Indirect costs - costs to the patient or family related to having the disease but not to direct health care.

   b. Out of pocket (OOP) - costs paid in cash or credit for health-related expenses not covered by the public health or private insurance systems.
2. Determine the sociodemographic and disease characteristics associated with higher costs

Methods:

Population: Incident cases of IBD (<16y) over 12 months (est. enrollment 250-300).

Indirect and OOP disease-related costs will be determined with surveys conducted one year following diagnosis and every 6mo for 2y. These will be conducted querying families on the preceding 4 weeks including: school and work days missed, out-of-pocket expenses, distance travelled to appointments, medications expenses incurred, and disability benefits collected. Indirect costs will be calculated using the Human Capital Approach (gross income not earned due to disease).

DETAILED DESCRIPTION:
Specific objectives:

1. Determine the Indirect and out of pocket costs of care of children with IBD, incurred by caregivers, funders, and the health system. Costs include:

   1. Indirect costs - all costs related to the patient having the disease but not related to direct health care costs. These include those paid by the patient, family, insurance system, and public funding. These include but are not limited to the costs of lost productivity hours due to missed work, missed school and volunteering activities, employment or disability insurance costs.
   2. Out of pocket (OOP) costs - those paid by the patient or family of the patient in cash or credit for healthcare related expenses that are not covered by the public health or insurance systems. These include but are not limited to medication dispensing fees, parking costs for medical appointments, travel expenses for medical appointments, special diet, alternative health treatments, and any other incurred disease-related costs such as educational books and donations.
2. Determine the sociodemographic and disease characteristics associated with higher costs

Background:

Inflammatory bowel disease (IBD) is a group of disorders characterized by chronic inflammation of the gastrointestinal tract with remissions and relapses. The two most common subtypes are Crohn's disease (CD) and ulcerative colitis (UC). The incidence of IBD appears to have risen over the last twenty years especially in the pediatric population.1-4 IBD is often diagnosed in the second or third decades of life, and therefore can impact both patients' social functioning and wellbeing, but also the family unit.. In addition, the fact that patients are most frequently diagnosed while in school or soon after, can result in significant cost to both the health system and to the economy. In 2012, the burden-of-illness report from the Crohn's and Colitis Canada estimated that the direct medical costs of IBD in Canada were over one billion dollars, primarily funded through the Canadian public healthcare system.1 While many international studies examined IBD-related costs in adults, information on direct and indirect health care costs resulting from a childhood diagnosis of IBD is not readily available.

Review of the Canadian Literature in Adult IBD: Members of our group investigated the direct hospital costs from the payer perspective for a cohort of 187 CD and 115 UC adult patients at a tertiary care hospital in Manitoba, in 1994-1995. The mean cost of hospital admission per medical case was C$2571 (95% CI, C$1801-C$3340) for CD and C$2186 (95% CI, C$1449-C$2922) for UC. The mean cost per hospitalized surgical case was higher, with C$3427 (95% CI, C$2728-C$4126) for CD and C$4635 (95% CI, C$3549-C$5726) for UC. Using the median values per hospitalized patient, the medical cost was C$1664 for CD and C$1262 for UC; the surgical cost was C$2546 for CD and C$3341 for UC. Surgery accounted for 50% of all hospital admissions, 58% of all hospital days, and 61% of all costs.5 The same investigators used administrative data to estimate health care utilization in adults with IBD in Manitoba. They concluded that the first 2 years from disease diagnosis were the most costly in terms of health care utilization.6 Longobardi et al examined indirect costs in the form of work loss related to IBD. Approximately 29% of adults with IBD reported labor force non-participation. The investigators estimated IBD-related indirect costs attributable to nonparticipation in 1998 to be over C$104 million.7 In another study from Manitoba, an acceptable concordance between patient-reported and administrative data-driven health care utilization.8 A high rate of concordance was also reported in a recent study from the Netherlands.9 This specific question of self-reported versus health records-reported health care utilization has never been examined in pediatric IBD.

A population-based surveillance cohort from Alberta examined predictors of costs for adults with UC who were hospitalized for a flare or colectomy between 2001 and 2009. Median hospitalization cost for UC flare, emergent colectomy and elective colectomy were: C$5,499, C$23,698 and C$14,316, respectively. Adjusted hospitalization costs increased approximately 6% annually. Use of infliximab was an independent predictor of increased costs.10 Economic data for a small adult sample hospitalized for Crohn's disease in Alberta, assessed costs two years before and after infliximab therapy. Total health care resource use and direct health care costs were compared for patients with or without fistulae. In the year following initiation of infliximab therapy, there were significant decreases in health care use, reflected in total hospital days, inpatient and outpatient colonoscopies and major surgeries.11 Review of Pediatric IBD Research: Using a collection of American HMO administrative data, Kappelman et al described the healthcare utilization and direct costs associated with IBD in insured American children and adults with IBD. Overall, healthcare utilization was higher in children with IBD compared to adults and in patients with CD compared to those with UC. Mean annual direct health costs for CD and UC were US$8,265 and US$5,066 respectively. In children, direct costs were approximately double that of .12 In a cross-sectional study Sin et al estimated the out of pocket (OOP) costs in parents of 150 children with IBD in California through surveys. Over 28% of those parents estimated their annual OOP costs to be more than US$1,000. Uncontrolled, severe, and frequently relapsing IBD correlated with higher OOP costs.13 In another retrospective cross-sectional analysis from Canterbury, New Zealand, the annual total costs per patient for pediatric CD were NZ$14,375 with direct and indirect costs comprising NZ$12,583 and NZ$1,792, respectively. Based on these data, the investigators estimated the annual total direct and indirect costs of CD across New Zealand to be approximately NZ$25.9 million.14 In a single center study, Wu et al, examined non-drug costs associated with outpatient infliximab infusions in children with IBD. The total annual drug cost was approximately $393,000 in 2011. For direct costs related to infliximab infusions, more than 77% of the total health care costs were related to personnel (e.g., nursing), facility operations, and laboratory costs. Only 23% of the total costs were related to the actual infliximab drug costs.15

Rationale:

In its 2012 report on the burden of IBD in Canada, Crohn's and Canada estimated that direct medical costs for IBD were C$1.2 billion, and that indirect costs were C$1.6 billion. Accordingly, the total annual costs for IBD in Canada were approximately C$2.8 billion. It is well-recognized that IBD causes significant financial burden on the economy, which is likely rising due to increased prevalence of the disease and the increasing use of high-cost biologic medications. Disease-related costs in Canadian children with IBD have never been studied. Therefore, we will conduct a national Canadian study examining IBD-related health costs, a crucial step to plan for proper allocation of resources and for future health services for Canadian children with IBD.

The cohort of recently developed CIHR/CHILD Foundation Canadian Children IBD Network (CIDsCaNN) includes about 1000 IBD patients. This network comprises 12 pediatric IBD centres across Canada tasked with the creation of an inception cohort of all children diagnosed with IBD. Biological and clinical information, including medication utilization, disease phenotype and disease severity is collected, with longitudinal follow-up.

Methods:

Source Population: Incident cases of pediatric IBD (<17y) in (CIDsCaNN) centres enrolled over a 12 month period or after (estimated enrollment 250-300 over a period of 12 months). Patients will be expected to be followed for a minimum of 2 years Study Design: A prospective cohort study will be conducted to determine disease-related costs using a series of cross-sectional surveys (Appendix). Surveys will be conducted at 6-18 months following the diagnosis then every 6 months for 2 years through the CIDsCaNN web portal, querying families on activity in the 4 weeks prior to the survey: school (patient) and work (parents) days missed, out-of-pocket expenses, distance travelled to care appointments, medications expenses incurred, and disability benefits collected. If participants are unable to complete the survey online, research assistant will give them the survey in a paper format to be completed.

Duration of costs covered: The survey will collect direct (6 months period), indirect and OOP costs in the 4 weeks preceding the survey (4 surveys over the study period) Indirect and OOP costs will be calculated in Canadian dollars, and adjusted for inflation using an appropriate inflationary measure (such as the Consumer Price Index (CPI)). Indirect costs will be calculated using the Human Capital Approach (gross income not earned due to disease).20 All costs will be adjusted for inflation using an inflationary measure such as CPI for health and personal care, by province (March 2016) 21.

Predictors of increased costs will be determined, with variables assessed to include: gender, age, pediatric IBD centre, family income, parents level of education, region of residence, disease duration, disease phenotype using Paris modification of Montreal classification, clinical activity at diagnosis and one year after diagnosis as measured by pediatric Crohn's activity index for CD (PCDAI) and pediatric UC activity index for UC (PUCAI), and adherence to IBD medications.

Statistical Analysis: Descriptive statistics will be reported as means with standard deviations (SD), medians with interquartile range (IQR), or proportions where appropriate. Two-part models will be estimated, in which the likelihood of incurring any expenditures and the natural logarithm of conditional expenditures will be estimated separately by logistic and ordinary least-squares models.

ELIGIBILITY:
Inclusion Criteria:

* Incident cases of pediatric IBD (<17y) in (CIDsCaNN) centres enrolled over a 12 month period (estimated enrollment 300-400 patients).

Exclusion Criteria:

* Non confirmed IBD

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Incident cases of pediatric IBD (<17y) in (CIDsCaNN) centres enrolled over a 12 month period (estimated enrollment 300-400 patients).
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-11-07 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Costs of care of children with IBD incurred by caregivers | 24 months
  Questionnaire: mean one month cost per patient in Canadian dollars

CONTACTS AND LOCATIONS:
Overall Officials: WAEL EL-MATARY, MD, Principal Investigator — Associate Professor, Section Head, Pediatric Gastroenterology
Locations (1):
- Winnipeg Children's Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] El-Matary W, Witt J, Bernstein CN, Jacobson K, Mack D, Otley A, Walters TD, Huynh HQ, deBruyn J, Griffiths AM, Benchimol EI. Indirect and Out-of-Pocket Disease-associated Costs in Pediatric Inflammatory Bowel Disease: A Cross-sectional Analysis. J Pediatr Gastroenterol Nutr. 2022 Oct 1;75(4):466-472. doi: 10.1097/MPG.0000000000003545. Epub 2022 Jun 27. PMID 35758424